CLINICAL TRIAL: NCT05151068
Title: Study on the Effect of Acupoint Application Combined With Ear Acupoint Embedding on the Discomfort Symptoms of Nasal Catheterization in Patients After Esophageal Cancer Surgery
Brief Title: the Effect of Acupoint Application Combined With Ear Acupoint Embedding in Patients After Esophageal Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210928
Record Dates: First submitted 2021-10-21; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Traditional Chinese Medicine
Keywords: acupoint application; ear acupoint embedding; esophageal cancer surgery; unplanned extubation; thirst; thore throat; comfort; sleep

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A,traditional (Experimental): The control group is given conventional nursing care: ①Preoperative education, informing patients of the importance of the tube and the adverse effects of unauthorised extubation after the operation on the recovery of the disease. ②Pipe care: The nose wing is fixed with modified "human" elastic tape, and the same side cheek bridge is fixed to keep the duct unobstructed and pour gastric juice in time. ③Oral care: routinely brush teeth and gargle with mouthwash daily. ④Skin care: Observe the condition of the nose, cheek skin and oral and nasal mucosa. Replace the tape as needed, and clean the skin before fixing. ⑤ Pain care: assess the degree of pain, follow the doctor's prescription for medication, and observe the efficacy of medication. ⑥Psychological care: pay attention to the emotional changes of patients and provide psychological support.This group is planned to enroll 100 patients.
  Interventions: Behavioral: traditional nursing method
- Group B,Precise (Experimental): On the basis of conventional nursing, the experimental group adopted a precision nursing program of acupoint application combined with ear acupoint embedding.This group is planned to enroll 100 patients.
  Interventions: Behavioral: Precise acupoint application combined with ear acupoint embedding nursing program

INTERVENTIONS:
Behavioral: traditional nursing method — ①Preoperative education, informing patients of the importance of the tube and the adverse effects of unauthorised extubation after the operation on the recovery of the disease. ②Pipe care: The nose wing is fixed with modified "human" elastic tape, and the same side cheek bridge is fixed to keep the duct unobstructed and pour gastric juice in time. ③Oral care: routinely brush teeth and gargle with mouthwash daily. ④Skin care: Observe the condition of the nose, cheek skin and oral and nasal mucosa. Replace the tape as needed, and clean the skin before fixing. ⑤ Pain care: assess the degree of pain, follow the doctor's prescription for medication, and observe the efficacy of medication. ⑥Psychological care: pay attention to the emotional changes of patients and provide psychological support.
  Arms: Group A,traditional
Behavioral: Precise acupoint application combined with ear acupoint embedding nursing program — On the basis of conventional nursing, the experimental group adopted a precision nursing program of acupoint application combined with ear acupoint embedding.
  Arms: Group B,Precise

SUMMARY:
To study the effect of acupoint application combined with ear acupoint seeding on the discomfort symptoms of nasal catheter in patients after esophageal cancer surgery

DETAILED DESCRIPTION:
From January to December 2021, 200 patients after esophageal cancer surgery with nasal catherterization in an affiliated hospital of Soochow will be selected as the research objects, and they will be divided into experimental group (100 cases) and control group (100 cases) by random number table method. The control group will receive routine nursing care, and the experimental group will implement a precision nursing program of acupoint application combined with ear acupoint embedding on the basis of the control group. The thirst, throat pain, comfort, sleep, and unplanned extubation rate will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Meet the diagnostic criteria for esophageal cancer; Age 50-70 years old; Undertake radical surgery for esophageal cancer, and place a tube through the nose after surgery; The patient communicates well with no cognitive impairment; Informed consent for this study, signed informed consent .

Exclusion Criteria:

Patients undergoing mechanical ventilation after surgery; Serious complications and death after surgery; Patients with external ear diseases and skin damage; Participating in other clinical research projects.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
unplanned extubation | Through study completion,an average of 7 days.
  Unplanned extubation refers to the early withdrawal of the catheter due to various reasons before the end of the treatment. This study includes the partial or complete extubation of the patient during the catheterization period. The calculation formula: (The number of cases of unplanned extubation in the group/the number of patients in the same group during the same period) × 100%.
The change of thirst | Evaluate at 12 hours, 24 hours, 48 hours, 72 hours and 7 days after surgery
  Thirst is assessed by the Visual Analogue Scale (VAS), and the higher the score, the more severe the patients' thirst .
The change of throe throat | Evaluate at 12 hours, 24 hours, 48 hours, 72 hours and 7 days after surgery
  Thore throat is evaluated by NRS. The higher the score, the more severe the throat pain of the patient.
The change of comfort | Evaluate at admission, 24 hours, 48 hours, 72 hours and 7 days.
  The comfort state is evaluated by Gnneral comfort questionnaire(GCQ). The scale includes 4 dimensions of physiology, psychology, spirit, social culture and environment, with a total of 28 items. The higher the score, the better the patient's comfort state.
The change of sleep | Evaluate at admission, 24 hours, 48 hours, 72 hours and 7 days.
  Sleep is evaluated using Athens insomnia scale (AIS). The higher the score, the worse the quality of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Luo, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The first affiliated hospital of soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang TR, Han Y, Liu B, Du MB, Xiang YH, Du XH, Li ZX, Jiao Y. [Observation of acupoint application of gel plaster on insomnia]. Zhongguo Zhen Jiu. 2021 May 12;41(5):505-9. doi: 10.13703/j.0255-2930.20200423-0005. Chinese. PMID 34002563
- [Background] Yuan J, Chen Y, Yu P, Luo F, Gao Y, Chen J, Wang P, Wang Y, Zhao Y, Lei Y. Effect of magnetic stimulation of Shenmen point on cognitive function of chronic insomnia: A randomized controlled clinical trial. Medicine (Baltimore). 2020 Dec 18;99(51):e23807. doi: 10.1097/MD.0000000000023807. PMID 33371157
- [Background] Ko YL, Lin SC, Lin PC. Effect of auricular acupressure for postpartum insomnia: an uncontrolled clinical trial. J Clin Nurs. 2016 Feb;25(3-4):332-9. doi: 10.1111/jocn.13053. Epub 2015 Nov 27. PMID 26612319
- [Background] Sun JL, Sung MS, Huang MY, Cheng GC, Lin CC. Effectiveness of acupressure for residents of long-term care facilities with insomnia: a randomized controlled trial. Int J Nurs Stud. 2010 Jul;47(7):798-805. doi: 10.1016/j.ijnurstu.2009.12.003. Epub 2010 Jan 6. PMID 20056221
- [Background] Fu HY, Chen QZ, Huang ZY, Wei CN. [Effect of auricular point pressing combined with electroacupuncture on postoperative pain and inflammatory cytokines in children with hernia]. Zhongguo Zhen Jiu. 2019 Jun 12;39(6):583-7. doi: 10.13703/j.0255-2930.2019.06.004. Chinese. PMID 31190492
- [Background] Long Q, Li Y, Li J, Wen Y, Du W, Wan C, Yue C. [Clinical observation of electroacupuncture combined with auricular point sticking therapy for anal pain of mixed hemorrhoid after external excision and internal ligation]. Zhongguo Zhen Jiu. 2018 Jun 12;38(6):580-5. doi: 10.13703/j.0255-2930.2018.06.003. Chinese. PMID 29971998
- [Background] Li L, Wang J, Li Y. [Effects of auricular plaster therapy on quality of life in uremia patients after parathyroidectomy plus autograft]. Zhongguo Zhen Jiu. 2017 Sep 12;37(9):938-43. doi: 10.13703/j.0255-2930.2017.09.007. Chinese. PMID 29354913
- [Background] Wang Z, Ma J, Ning L. [Clinical observation of dysphagia after cerebral infarction treated with awn-like needle at Tiantu(CV 22)]. Zhongguo Zhen Jiu. 2016 Oct 12;36(10):1019-1022. doi: 10.13703/j.0255-2930.2016.10.004. Chinese. PMID 29231518